CLINICAL TRIAL: NCT01241942
Title: Phase 2 Study of Ex-vivo Perfusion and Ventilation of Lungs to Assess Transplant Suitability
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding exhausted.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Vitrolife (Industry); XVIVO Perfusion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: UNC-001 Vitrolife
Record Dates: First submitted 2010-11-12; First posted 2010-11-16 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Emphysema; Chronic Obstructive Pulmonary Disease (COPD); Cystic Fibrosis; Pulmonary Fibrosis; Bronchiectasis; Sarcoidosis; Pulmonary Hypertension; Alpha-1 Antitrypsin Deficiency
Keywords: Lung Transplant; Emphysema; Chronic Obstructive Pulmonary Disease (COPD); Cystic Fibrosis; Pulmonary Fibrosis; Bronchiectasis; Sarcoidosis; Pulmonary Hypertension; Alpha-1 Antitrypsin Deficiency
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive; Cystic Fibrosis; Pulmonary Fibrosis; Bronchiectasis; Sarcoidosis; Hypertension, Pulmonary; alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- EVLP with STEEN Solution™ (Experimental): The perfusion of the lungs will be performed using STEEN Solution™ and then physiologically assessed. Lungs deemed suitable will be transplanted after Ex-vivo Perfusion w/ STEEN Solution™.
  Interventions: Device: Steen Solution™
- Conventional Lung transplant (Active Comparator): No experimental procedures will be carried out. Lungs from conventional brain-dead organ donors will be used for transplant.
  Interventions: Other: Conventional Lung Transplant

INTERVENTIONS:
Device: Steen Solution™ — This solution is a buffered dextran and albumin-containing extracellular perfusate with an optimal colloid osmotic pressure developed specifically for extra-corporeal perfusion of lungs. After EVLP, lungs will be cooled in the circuit to room temperature, then flushed with cold Perfadex™ and taken to UNC Hospitals (UNCH) where they will have an ex-vivo CT scan. Lungs determined suitable will be offered to consented patients at UNCH based on Lung Allocation Score. Lungs not considered for transplantation may be subjected to different experiments but are not to be a part of this research study. In summary, lungs with good and stable function during EVLP with Steen Solution™ will be transplanted into recipients as per current clinical practice.
  Arms: EVLP with STEEN Solution™
Other: Conventional Lung Transplant — No experimental procedures will be carried out. Lungs from conventional brain-dead organ donors will be used for transplant.
  Arms: Conventional Lung transplant

SUMMARY:
The purpose of this research study is to perfect the technique of EVLP and learn about the safety of transplanting lungs that have been ventilated (attached to a breathing machine or ventilator to deliver oxygen) and perfused with a lung perfusion solution (Steen solution™, made by Vitrolife). This ventilation and perfusion will be done outside the body (ex-vivo) in a modified cardiopulmonary bypass circuit (the kind of device used routinely during most heart surgeries). The purpose of performing ex-vivo lung perfusion and ventilation (EVLP) is to learn how well the lungs work, and whether they are likely safe to transplant.

ELIGIBILITY:
Lung Recipient Inclusion Criteria:

* A recipient must meet the following requirement to enroll into the study:
* Requires a single or bilateral lung transplant and is listed for lung transplant at UNC.
* Male or Female, 18 years of age or older.
* Subject or Subject's Representative provides a legally effective informed consent.
* Recipient does not have HIV, active Hepatitis or is colonized with Burkholderia cepacia.
* Potential subjects who have undergone previous lung transplants and meet all other inclusion criteria are eligible for study participation.

Lung Recipient Exclusion Criteria:

* Recipient fails to meet standard of care requirements for lung transplant, or decides not to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
30 Day Mortality | 30 Days
  The primary objective evaluated for this study is recipient mortality at 30 days post transplant. 30 day mortality is used as a standard research assessment to evaluate post transplant outcomes.

SECONDARY OUTCOMES:
Primary Lung Graft Dysfunction (PGD) | 24 and 72 hours post transplant.
  Primary Lung Graft Dysfunction (PGD) is an indicator for significant morbidity and mortality after lung transplantation.
  Grade 0: PaO2*/FIO2** > 300 with normal chest radiograph; Grade 1: PaO2/FIO2 > 300 with diffuse infiltrates on the chest radiograph; Grade 2: PaO2/FIO2 between 200 and 300; Grade 3: PaO2/FIO2 < 200.
  * partial pressure of oxygen in the arterial blood (PaO2)
  ** fraction of inspired oxygen inspired oxygen fraction (FIO2)
ICU Length of Stay | Time to Discharge.
  The length of ICU stay is another standard research and clinical outcome assessment post transplant and has been selected as a secondary objective.
Day 7 Ventilator/ECMO Status | 7 Days Post Transplant.
  7 days ventilator or extra-corporeal membrane oxygenator (ECMO free are being evaluated as secondary objectives.
Recipient mortality at 12 months. | 12 months
  Recipient mortality at 12 months post transplant is being evaluated as a secondary objective.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M. Egan, MD, MSc., Principal Investigator — UNC-Chapel Hill
Locations (1):
- UNC Hospitals, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Orens JB, Estenne M, Arcasoy S, Conte JV, Corris P, Egan JJ, Egan T, Keshavjee S, Knoop C, Kotloff R, Martinez FJ, Nathan S, Palmer S, Patterson A, Singer L, Snell G, Studer S, Vachiery JL, Glanville AR; Pulmonary Scientific Council of the International Society for Heart and Lung Transplantation. International guidelines for the selection of lung transplant candidates: 2006 update--a consensus report from the Pulmonary Scientific Council of the International Society for Heart and Lung Transplantation. J Heart Lung Transplant. 2006 Jul;25(7):745-55. doi: 10.1016/j.healun.2006.03.011. No abstract available. PMID 16818116
- [Background] Ingemansson R, Eyjolfsson A, Mared L, Pierre L, Algotsson L, Ekmehag B, Gustafsson R, Johnsson P, Koul B, Lindstedt S, Luhrs C, Sjoberg T, Steen S. Clinical transplantation of initially rejected donor lungs after reconditioning ex vivo. Ann Thorac Surg. 2009 Jan;87(1):255-60. doi: 10.1016/j.athoracsur.2008.09.049. PMID 19101308
- [Background] Mason DP, Thuita L, Alster JM, Murthy SC, Budev MM, Mehta AC, Pettersson GB, Blackstone EH. Should lung transplantation be performed using donation after cardiac death? The United States experience. J Thorac Cardiovasc Surg. 2008 Oct;136(4):1061-6. doi: 10.1016/j.jtcvs.2008.04.023. PMID 18954650
- [Background] Cypel M, Yeung JC, Hirayama S, Rubacha M, Fischer S, Anraku M, Sato M, Harwood S, Pierre A, Waddell TK, de Perrot M, Liu M, Keshavjee S. Technique for prolonged normothermic ex vivo lung perfusion. J Heart Lung Transplant. 2008 Dec;27(12):1319-25. doi: 10.1016/j.healun.2008.09.003. PMID 19059112
- [Background] Egan TM, Haithcock JA, Nicotra WA, Koukoulis G, Inokawa H, Sevala M, Molina PL, Funkhouser WK, Mattice BJ. Ex vivo evaluation of human lungs for transplant suitability. Ann Thorac Surg. 2006 Apr;81(4):1205-13. doi: 10.1016/j.athoracsur.2005.09.034. PMID 16564244
- [Background] Christie JD, Carby M, Bag R, Corris P, Hertz M, Weill D; ISHLT Working Group on Primary Lung Graft Dysfunction. Report of the ISHLT Working Group on Primary Lung Graft Dysfunction part II: definition. A consensus statement of the International Society for Heart and Lung Transplantation. J Heart Lung Transplant. 2005 Oct;24(10):1454-9. doi: 10.1016/j.healun.2004.11.049. Epub 2005 Jun 4. No abstract available. PMID 16210116
- [Background] Kim IK, Bedi DS, Denecke C, Ge X, Tullius SG. Impact of innate and adaptive immunity on rejection and tolerance. Transplantation. 2008 Oct 15;86(7):889-94. doi: 10.1097/TP.0b013e318186ac4a. PMID 18852649
- [Background] Moers C, Smits JM, Maathuis MH, Treckmann J, van Gelder F, Napieralski BP, van Kasterop-Kutz M, van der Heide JJ, Squifflet JP, van Heurn E, Kirste GR, Rahmel A, Leuvenink HG, Paul A, Pirenne J, Ploeg RJ. Machine perfusion or cold storage in deceased-donor kidney transplantation. N Engl J Med. 2009 Jan 1;360(1):7-19. doi: 10.1056/NEJMoa0802289. PMID 19118301
- [Background] Cypel M, Liu M, Rubacha M, Yeung JC, Hirayama S, Anraku M, Sato M, Medin J, Davidson BL, de Perrot M, Waddell TK, Slutsky AS, Keshavjee S. Functional repair of human donor lungs by IL-10 gene therapy. Sci Transl Med. 2009 Oct 28;1(4):4ra9. doi: 10.1126/scitranslmed.3000266. PMID 20368171
- See also: Organ Procurement and Transplantation Network web site (National Data/ Waiting List Removals/ Lung/ Removal Reasons by Year) — https://optn.transplant.hrsa.gov/